CLINICAL TRIAL: NCT06649370
Title: Effect of Systemic Inflammatory Index and Systemic Immune Inflammation Index on Ecchymosis, Bleeding and Edema in Rhinoplasty.
Brief Title: Effect of Systemic Inflammatory Index and Systemic Immune Inflammation Index on Ecchymosis, Bleeding and Edema
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 24-KAEK-185
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Rhinoplasty
Keywords: Ecchymosis; Edema; Inflammation; Platelet Count
MeSH Terms: conditions — Ecchymosis; Edema; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Hypotensive Drugs and/or Vasoactive Drugs — If the patients' mean arterial pressure falls below 60 mmHg or 20% below the preoperative value, ephedrine will be administered.

SUMMARY:
Rhinoplasty is a cosmetic surgical procedure that is widely applied today and is characterized by edema in the postoperative period. In particular, edema can cause prolonged recovery and deterioration in the patient's social life. Various studies have been conducted using certain drugs or different surgical techniques to reduce edema and ecchymosis in rhinoplasty.

In rhinoplasty, edema occurs after the absorption of interstitial fluid in the nose is disrupted as a result of trauma to the bone and soft tissue. Ecchymosis occurs when blood passes from damaged vessels due to surgery to the loose and thin soft tissue around the eye. Ecchymosis is often seen on the eyelids after open rhinoplasty. Ecchymosis usually moves in the direction of gravity and increases in the first two days after surgery.

Systemic inflammatory response index and systemic immune inflammation index can be easily obtained with a simple hemogram test. These indexes have been suggested to be a useful parameter in many diseases associated with inflammation, but research is still ongoing. Inflammation values and the resulting response have an important effect on wound formation and healing. However, increased inflammation can also increase edema and ecchymosis in the postoperative period. In this study, the researchers aimed to investigate the relationship between preoperative inflammation values and postoperative edema and ecchymosis in open rhinoplasties.

DETAILED DESCRIPTION:
Although rhinoplasty is one of the most commonly performed facial surgical procedures, intraoperative bleeding, postoperative ecchymosis and edema negatively affect patient satisfaction. No matter how gently and carefully the surgeon performs the procedure in rhinoplasty, trauma, inflammation and as a result edema and ecchymosis develop in the tissues. Edema and ecchymosis can cause temporary vision loss, permanent pigmentation and scar tissue. Studies have been conducted using different drugs such as steroids, adrenaline and lidocaine to reduce edema and ecchymosis in rhinoplasty surgery and different osteotomy techniques in rhinoplasty. In patients undergoing rhinoplasty, inflammation of the nasal mucosa at the osteotomy site is an important cause of periorbital edema and ecchymosis. The systemic inflammatory response index is an easily accessible and calculable biomarker that provides important information about inflammatory conditions and inflammatory diseases. This simple index shows the balance between regulatory and protective lymphocytes, neutrophils and active inflammatory components. In addition to inflammation, this index also provides information about vascular involvement and damage in some diseases. Leukocytes further increase inflammation in damaged vessels, increasing endothelial damage and the risk of thrombus. Rhinoplasty is a commonly performed surgical procedure, and postoperatively, even during the surgical procedure, ecchymosis and edema can be seen around the eyes and face. This affects the patient's recovery, discharge, and return to social life. Many studies have been conducted to reduce postoperative edema and ecchymosis in rhinoplasty. However, it is very important to be able to predict the severity of edema and ecchymosis in advance. There are not enough studies on this subject, and the results are contradictory. Therefore, the aim of this study was to investigate whether there is a relationship between the systemic inflammatory response index and systemic immune inflammation index, which are measured before surgery in rhinoplasty, and postoperative ecchymosis and edema.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planning to undergo rhinoplasty and are between the ages of 18-45 are willing to participate in the study.

Exclusion Criteria:

* Heart failure
* Severe respiratory failure
* Renal failure
* Vascular diseases
* Steroid use
* Coagulation disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective, randomized, controlled observational study will be conducted on patients undergoing open rhinoplasty with osteotomy. Rhinoplasty patients aged 18-45 years who will undergo general anesthesia and have an American Society of Anesthesiologists (ASA) score of 1 and 2 will be included in the study.
  The sample size was calculated with a type 1 error value of 0.05, a power of 0.80 and r = 0.30 (low-level correlation) between the systemic inflammatory index and edema score, and 85 patients were considered sufficient for the study. Considering the losses that may occur during follow-up, it was planned to conduct the study with 94 patients with a 10% increase.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
postoperative edema and ecchymosis | Each patient will be evaluated on postoperative days 1, 2 and 7.
  Each patient will be photographed with a digital camera on postoperative days 1, 2, and 7. Eyelid edema and periorbital soft tissue ecchymosis will be assessed using a separate grading scale (range 0-4). The assessment will be performed by an independent observer for each patient on the indicated days.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided